CLINICAL TRIAL: NCT04400331
Title: Open-Label Rollover Study for Continuing Valbenazine Administration for the Treatment of Chorea Associated With Huntington Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Huntington Study Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-HD3006
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Chorea, Huntington
MeSH Terms: conditions — Huntington Disease | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valbenazine (Experimental): Capsule, administered orally once daily.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: NBI-98854

SUMMARY:
This is a Phase 3, open-label study to evaluate the long-term safety and tolerability of valbenazine, and to provide participants continued access to valbenazine for the treatment of chorea associated with Huntington disease.

DETAILED DESCRIPTION:
After completion of Week 156/early termination visit, participants in the US will be given the option to continue into an extended maintenance period for up to 104 weeks and participants in Canada will have the option to participate in a separate open-label study (Study NBI-98854-HD3022).

ELIGIBILITY:
Inclusion Criteria:

Either #1 or #2 must be met for inclusion eligibility.

1. Have participated in Study NBI-98854-HD3005 and

   a. Study drug dosing completion of Study NBI-98854-HD3005, as demonstrated by completed study drug dosing through the follow-up visit or early terminated Study NBI-98854-HD3005 for administrative reasons due to COVID-19 (for example, site closure related to COVID-19)
2. Did not participate in Study NBI-98854-HD3005 and

   1. Have a clinical and genetic diagnosis of Huntington Disease (HD) with chorea
   2. Be able to walk, with or without the assistance of a person or device
3. Be able to read and understand English and capable of providing consent to study participation or have a legally authorized representative providing consent and the participant providing assent
4. Participants of childbearing potential must agree to use contraception consistently while participating in the study until 30 days after last dose of the study treatment

Exclusion Criteria:

1. Have difficulty swallowing
2. Are currently pregnant or breastfeeding
3. Have a known history of long QT syndrome, cardiac tachyarrhythmia, left bundle-branch block, atrioventricular (AV) block, uncontrolled bradyarrhythmia, or heart failure
4. Have an unstable or serious medical or psychiatric illness
5. Have a significant risk of suicidal behavior
6. Have a history of substance dependence or substance (drug) or alcohol abuse, within 1 year of screening
7. Have received gene therapy at any time
8. Have received an investigational drug in a clinical study (other than valbenazine) within 30 days before the baseline visit or plan to use such investigational drug (other than valbenazine) during the study
9. Have had a blood loss ≥550 mL or donated blood within 30 days before the baseline visit
10. Have a history of severe hepatic impairment or history of protocol specified hematologic abnormalities during the course of the NBI-98854-HD3005 study
11. Had a medically significant illness within 30 days before baseline, or any history of neuroleptic malignant syndrome
12. Have a known hypersensitivity to any component of the formulation of valbenazine
13. For participants who did not participate in NBI-98854-HD3005: have a history of VMAT2 inhibitor use within 30 days of baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 262 weeks

SECONDARY OUTCOMES:
Change from Baseline in the Unified Huntington's Disease Rating Scale (UHDRS) Total Maximal Chorea (TMC) Score | Up to 262 weeks
  The TMC is part of the motor assessment of the UHDRS and measures chorea in 7 different body parts including the face, oral-buccal-lingual region, trunk and each limb independently. The TMC score is the sum of the individual scores and ranges from 0 to 28. A decrease in score indicates improvement in chorea.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Chief Medical Officer
Locations (33):
- United States (30):
  - Neurocrine Clinical Site, Birmingham, Alabama
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, La Jolla, California
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Washington D.C., District of Columbia
  - Neurocrine Clinical Site, Boca Raton, Florida
  - Neurocrine Clinical Site, Gainesville, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Indianapolis, Indiana
  - Neurocrine Clinical Site, Iowa City, Iowa
  - Neurocrine Clinical Site, Wichita, Kansas
  - Neurocrine Clinical Site, Louisville, Kentucky
  - Neurocrine Clinical Site, New Orleans, Louisiana
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Charlestown, Massachusetts
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Omaha, Nebraska
  - Neurocrine Clinical Site, Rochester, New York
  - Neurocrine Clinical Site, Williamsville, New York
  - Neurocrine Clinical Site, Durham, North Carolina
  - Neurocrine Clinical Site, Columbus, Ohio
  - Neurocrine Clinical Site, Toledo, Ohio
  - Neurocrine Clinical Site, Pittsburgh, Pennsylvania
  - Neurocrine Clinical Site, Charleston, South Carolina
  - Neurocrine Clinical Site, Columbia, South Carolina
  - Neurocrine Clinical Site, Greenville, South Carolina
  - Neurocrine Clinical Site, Nashville, Tennessee
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Burlington, Vermont
- Canada (3):
  - Neurocrine Clinical Site, Vancouver, British Columbia
  - Neurocrine Clinical Site, Ottawa, Ontario
  - Neurocrine Clinical Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://huntingtonstudygroup.org/current-clinical-trials/kinect-hd2/